CLINICAL TRIAL: NCT03983174
Title: Drainage Seton Around the External Anal Sphincter With Mucosal Advancement Flap Versus External Anal Sphincter Preserving Seton in Treatment of Trans-sphincteric Anal Fistula
Brief Title: Drainage Seton With Flap Versus EAS Preserving Seton in Treatment of Transsphincteric Anal Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mansoura102
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms | interventions — Surgical Flaps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drainage seton with flap (Experimental): Drainage seton will be put around the external anal sphincter with mucosal advancement flap
  Interventions: Procedure: Drainage seton with flap
- EAS sparing seton (Experimental): Rerouting of the seton around the internal anal sphincter sparing the external sphincter will be done
  Interventions: Procedure: EAS sparing seton

INTERVENTIONS:
Procedure: Drainage seton with flap — Seton is placed around the external sphincter then mucosal advancement flap will be constructed
  Arms: Drainage seton with flap
Procedure: EAS sparing seton — Rerouting of the seton around the internal sphincter only sparing the external sphincter
  Arms: EAS sparing seton

SUMMARY:
Patients with high trans-sphincteric anal fistula will be randomized to one of two equal group: group 1 will have drainage seton with mucosal advancement flap and group 2 will undergo external anal sphincter sparing seton

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from high trans-sphincteric anal fistula

Exclusion Criteria:

* Acute sepsis.
* Specific cause of fistula e.g. Crohn's disease
* Strictured anorectum.
* Any degree of incontinence
* Recurrent anal fistula.
* Low anal fistula.
* Previous anorectal surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
fecal incontinence | 12 months after surgery
  Number of patients who develop fecal incontinence as assessed by Wexner Incontinence score

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No